CLINICAL TRIAL: NCT02202616
Title: Prospective Cohort Study for the Real - Life Effectiveness Evaluation of GlycOpyrronium With IndacatERol Combination in the Management of COPD in Canada (POWER Study)
Acronym: POWER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQVA149ACA01
Record Dates: First submitted 2014-06-26; First posted 2014-07-29 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD,; QVA149,; Tiotropium,; FDC,; GlycOpyrronium With IndacatERol,; POWER
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ULTIBRO BREEZHALER (Other): Patients diagnosed with chronic obstructive pulmonary disorder (COPD) who are symptomatic (CAT score over 10) and who are treated with Tiotropium (SPIRIVA HANDALER) or Fluticasone propionate/Salmeterol- ADVAIR DISKUS (FDC).
  Interventions: Drug: Glycopyrronium /Indacaterol maleate

INTERVENTIONS:
Drug: Glycopyrronium /Indacaterol maleate — Glycopyrronium 50mcg/Indacaterol maleate 110mcg once daily by a breezhaler device

SUMMARY:
This is a single cohort, prospective post approval study conducted on patients with COPD in Canada. The study will enroll patients that have not responded to their current treatment of tiotropium alone, or who are on the fixed dose combinations fluticasone propionate/salmeterol. Only patients for whom the physician has decided to change treatment due to lack of efficacy will be eligible to be enrolled in the study.

Also will evaluate the real-life effectiveness of QVA149 (indacaterol 110 mcg/glycopyrronium 50 mcg) in the management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed and treated for moderate to severe COPD according to the Global Initiative for Chronic Obstructive Lung Disease according to physician's assessment
* Smoking history of > 10 pack - years.
* On-going treatment with tiotropium or fixed dose combination of LABA/ICS, specifically combinations fluticasone propionate/salmeterol for a minimum of three months but demonstrating persistence of symptoms indicating change of treatment to combination therapy **using a CAT score > 10.
* Treatment with QVA149 is indicated as per the product monograph and appropriate for the patient as per the judgment of the treating physician.
* Patient has signed informed consent agreeing to participate in the study and undergo the study treatments and allowing the use of their data for the purposes of the study.
* Patient is expected to be available for 16 weeks after study enrolment

  * Assessed as per routine care or as documented in the patient's chart. ** As determined and decided by the treating physician prior to enrolment of the patient in the study.

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study. No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible patients.

* Patients not willing to sign an informed consent.
* Patient on maintenance treatment including triple therapy (LABA +LAMA+ICS) for COPD
* Patients with a diagnosis of asthma or history of asthma.
* Patients who have had two or more moderate to severe exacerbations during the last 12 months prior to study enrolment. A moderate COPD exacerbation is defined by requirement for treatment with systemic corticosteroids or antibiotics or both. A severe COPD exacerbation is defined by hospitalization, including an emergency room visit of longer than 24 h.
* Patients who had an exacerbation within the previous 6 weeks to enrolment.
* Patients who as per physician clinical judgment will require ICS treatment co-administered with QVA149 during the study period.
* Patients with other chronic respiratory conditions that may affect the outcome of treatment including but not limited to lung cancer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Saint-Charles-Borromée, Quebec, Canada

REFERENCES:
- [Derived] Kaplan A, Chapman KR, Anees SM, Mayers I, Rochdi D, Djandji M, Prefontaine D, McIvor A. Real-life effectiveness of indacaterol-glycopyrronium after switching from tiotropium or salmeterol/fluticasone therapy in patients with symptomatic COPD: the POWER study. Int J Chron Obstruct Pulmon Dis. 2019 Jan 18;14:249-260. doi: 10.2147/COPD.S185485. eCollection 2019. PMID 30718952

RESULTS

PARTICIPANT FLOW:
Groups:
- QVA149 110/50: QVA149 110/50- Patients diagnosed with chronic obstructive pulmonary disorder (COPD) who are symptomatic (CAT score over 10) and who are treated with Tiotropium (SPIRIVA HANDALER) or Fluticasone propionate/Salmeterol- ADVAIR DISKUS (FDC).
Period: Overall Study
Arm/Group | QVA149 110/50
Started | 401
Intent to Treat Set (ITT) | 338
Completed | 301
Not Completed | 100
Not completed — Screen failed | 24
Not completed — Adverse Event | 32
Not completed — Protocol deviation | 18
Not completed — Patient withdrew consent | 12
Not completed — Lost to Follow-up | 6
Not completed — Administrative problems | 6
Not completed — Abnormal test procedure result | 1
Not completed — Unsatisfactory therapeutic effect | 1

BASELINE CHARACTERISTICS:
Population: The ITT included all patients who received the study treatment and returned for ≥ 1 post baseline visit
Arm/Group | ULTIBRO BREEZHALER
Number analyzed (Participants) | 338
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 189
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 330
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough (Forced Expiratory Volume (FEV1) (Pre-dose FEV1)
Description: Primary end points: To evaluate the real-life effectiveness of QVA149 (indacaterol 110 mcg/glycopyrronium 50 mcg) in the management of patients with COPD who have symptoms defined as CAT score >10 with tiotropium monotherapy; effectiveness will be assessed as the mean change in trough FEV1 from baseline to 16 weeks. and to evaluate the real-life effectiveness of QVA149 (indacaterol 110 mcg/glycopyrronium 50 mcg) in the management of patients with COPD who have symptoms defined as CAT score >10 while on treatment with FDC of fluticasone propionate/salmeterol; effectiveness will be assessed as the mean change in trough FEV1 from baseline to 16 weeks.
Time Frame: 16 weeks study
Population: Intent to treat set (ITT)- included all patients who received the study treatment and returned for ≥ 1 post baseline visit
Measure: Mean (Standard Deviation); unit: Liter
Groups:
- QVA149 110/50 After Flu/Sal: QVA149 110/50 combination of (indacaterol maleate 110 µg and glycopyrronium bromide 50 µg) after patients treated with FDC of fluticasone propionate and salmeterol
- QVA149 110/50 After Tio: QVA149 110/50 combination of (indacaterol maleate 110 µg and glycopyrronium bromide 50 µg) after patients treated with tiotropium
Arm/Group | QVA149 110/50 After Flu/Sal | QVA149 110/50 After Tio
Number analyzed (Participants) | 83 | 235
Liter | 0.17 (0.397) | 0.18 (0.321)
Statistical Analysis 1: Comparison: QVA149 110/50 After Flu/Sal vs QVA149 110/50 After Tio; Test type: Other; Descriptive Statistics with 95% CI; The mean change from baseline along with the 95% confidence interval used to assess the precision of the estimate; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.14 to 0.21], Standard Deviation 0.340

2. Secondary Outcome: Change From Baseline in Trough FEV1 (Forced Expiratory Volume) to Week 4
Description: Portable spirometers will be provided to investigators and they will use this device for all of their patient measurements of FEV1 during the trial
Time Frame: Baseline, week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | QVA149 110/50 After Flu/Sal | QVA149 110/50 After Tio
Number analyzed (Participants) | 79 | 224
Liter | 0.12 (0.308) | 0.14 (0.267)
Statistical Analysis 1: Comparison: QVA149 110/50 After Flu/Sal vs QVA149 110/50 After Tio; Test type: Other; Descriptive Statistics with 95% CI; The mean change from baseline along with the 95% confidence interval used to assess the precision of the estimate; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.11 to 0.17], Standard Deviation 0.278

3. Secondary Outcome: Single Point and Change in Baseline Dyspnea Index and Transitional Dyspnea Index (BDI/TDI)
Description: A trained assessor interviewed the patient and graded the degree of impairment due to dyspnea (difficulty breathing). BDI/TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort and captures changes from baseline. BDI was measured at day 1 prior to the first dose with domain scores ranging from 0=very severe to 4=no impairment and a total score ranging from 0 to 12(best). TDI captures changes from baseline. Each domain is scored from -3=major deterioration to 3=major improvement to give an overall TDI focal score of -9 to 9. Higher numbers indicate a better score. The BDI was assessed at Baseline, whereas the TDI was assessed at Week 4 and Week 16.
Time Frame: Baseline, Week 4, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | QVA149 110/50 After Flu/Sal | QVA149 110/50 After Tio
Number analyzed (Participants) | 87 | 248
Score
  BDI week 0: number analyzed (Participants) | 86 | 245
  BDI week 0 | 6.5 (2.07) | 6.8 (2.09)
  TDI week 4: number analyzed (Participants) | 79 | 226
  TDI week 4 | 2.2 (2.72) | 2.0 (2.38)
  TDI week 16: number analyzed (Participants) | 84 | 237
  TDI week 16 | 2.9 (3.28) | 2.4 (2.78)
Statistical Analysis 1: Comparison: QVA149 110/50 After Flu/Sal vs QVA149 110/50 After Tio; Week 4; Test type: Other; Standard Descriptive Statistics; The estimated mean change from baseline and corresponding 95% confidence intervals will be displayed for each visit; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [1.74 to 2.30], Standard Deviation 2.47
Statistical Analysis 2: Comparison: QVA149 110/50 After Flu/Sal vs QVA149 110/50 After Tio; Week 16; Test type: Other; Standard Descriptive Statistics; The estimated mean change from baseline and corresponding 95% confidence intervals will be displayed for each visit; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [2.21 to 2.85], Standard Deviation 2.92

4. Secondary Outcome: Change From Baseline in Chronic Obstructive Pulmonary Disease (COPD) Assessment Questionnaire (CAT)
Description: The CAT is an 8 item questionnaire that assesses the impact of COPD on the patient's functional status. Scores for each of the 8 items are summed to give an overall score (out of 40). The score ranges from 0-40 where higher scores represent worse health status. CAT scores ≥ 10 are associated with significantly impaired health status.
Time Frame: Baseline, week 4, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | QVA149 110/50 After Flu/Sal | QVA149 110/50 After Tio
Number analyzed (Participants) | 83 | 234
Score
  Week 4 | -5.9 (7.55) | -4.7 (5.71)
  Week 16 | -8.2 (8.34) | -5.9 (6.44)
Statistical Analysis 1: Comparison: QVA149 110/50 After Flu/Sal vs QVA149 110/50 After Tio; Week 4; Test type: Other; standard descriptive statistics; The estimated mean change from baseline to Week 4 along with the 95% confidence interval; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-5.7 to -4.3], Standard Deviation 6.25
Statistical Analysis 2: Comparison: QVA149 110/50 After Flu/Sal vs QVA149 110/50 After Tio; Week 16; Test type: Other; standard descriptive statistics; The estimated mean change from baseline to Week 4 along with the 95% confidence interval; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-7.3 to -5.7], Standard Deviation 7.03

ADVERSE EVENTS:
Time Frame: From week 0 to week 16
Groups:
- QVA149 110/50: QVA149 110/50-Patients diagnosed with chronic obstructive pulmonary disorder (COPD) who are symptomatic (CAT score over 10) and who are treated with Tiotropium (SPIRIVA HANDALER) or Fluticasone propionate/Salmeterol- ADVAIR DISKUS (FDC).
Arm/Group | QVA149 110/50
All-Cause Mortality (participants affected / at risk) | 0/373
Serious Adverse Events (participants affected / at risk) | 12/373
Other Adverse Events (participants affected / at risk) | 56/373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 110/50 (N=373)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Wound (Injury, poisoning and procedural complications) | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 110/50 (N=373)
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Bronchitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 11
Dizziness (Nervous system disorders) | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2015-06-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT02202616/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT02202616/SAP_001.pdf